CLINICAL TRIAL: NCT07063732
Title: The Effect of Ketone Monoester Supplementation and High Altitude on Exercising Cerebral Blood Flow
Brief Title: Ketone Monoester Supplements, High Altitude, and Brain Blood Flow During Exercise
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Jeremy Walsh, Assistant Professor, McMaster University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: KETEX_WM
Record Dates: First submitted 2025-05-28; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: High Altitude Hypoxia; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Altitude (3800m; Barcroft Research Station) (Experimental): High altitude setting
  Interventions: Dietary Supplement: Ketone Monoester (KME); Dietary Supplement: Placebo
- Low Altitude (334m; University of Guelph) (Experimental): Low altitude setting
  Interventions: Dietary Supplement: Ketone Monoester (KME); Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ketone Monoester (KME) — 0.6 g KME per kg body mass; [R]-3-hydroxybutyl [R]-3-hydroxybutyrate. (Delta G Ketone, TΔS, Oxford).
Dietary Supplement: Placebo — Inert, calorie-free placebo drink that is taste-matched to the ketone monoester supplement

SUMMARY:
The purpose of this trial is to investigate the effect of acute ketone monoester ingestion (0.6 g KME/kg body weight) on the occurrence of the ventilatory threshold and the subsequent response of blood velocity in cerebral arteries during a maximal exercise test at low altitude and high altitude.

ELIGIBILITY:
Inclusion Criteria:

- Must be a member of the research expedition team travelling to the Barcroft Research Station in White Mountain California

Exclusion Criteria:

* BMI > 30
* No prescribed medications (oral contraceptives excluded)
* History of smoking
* Currently following a ketogenic diet or consuming exogenous ketogenic supplements
* History of heart, lung, blood vessel, or kidney disease
* Currently pregnant

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Cerebral Blood Velocity | 3 hours
  Transcranial Doppler ultrasound will be used to measure blood velocity in the middle cerebral artery and posterior cerebral artery. Location of measurements will remain consistent within participants.

SECONDARY OUTCOMES:
Cardiac Output | 3 hours
  Cardiac output (L/min) will be measured using a non-invasive cardiac output monitor (Physioflow). The monitor uses signal morphology impedance cardiography to determine cardiac output.
Blood Pressure | 3 hours
  Mean arterial pressure (mmHg) will be measured via a brachial cuff placed on the upper arm.
Ventilatory Threshold | 3 hours
  Ventilatory threshold (VT) will be calculated based on previously described methods (Gaskill et al., 2001).
End-Tidal Gases | 3 hours
  End-tidal oxygen (PETO2) (mmHg) and carbon dioxide (PETCO2) (mmHg) will be collected using a metabolic cart.
Rate of Oxygen Consumption and Carbon Dioxide Production | 3 hours
  Rate of oxygen consumption (VO2) (mL/min) and carbon dioxide production (VCO2) (mL/min) will be collected using a metabolic cart.
Ventilation | 3 hours
  Ventilation (Ve) (L/min) will be collected using a metabolic cart.
Blood Lactate and Beta-Hydroxybutyrate | 3 hours
  Capillary blood will be obtained via finger prick using a lancing device to measure concentrations of blood lactate (mmol/L) and beta-hydroxybutyrate (mmol/L) using a handheld metabolite analyzer.
Peak Work Rate (Maximal Exercise Test) | 3 hours
  The maximum wattage (W) achieved by the participant during the maximal exercise test will be recorded.

CONTACTS AND LOCATIONS:
Locations (2):
- Barcroft Research Station, Bishop, California, United States
- University of Guelph, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gaskill SE, Ruby BC, Walker AJ, Sanchez OA, Serfass RC, Leon AS. Validity and reliability of combining three methods to determine ventilatory threshold. Med Sci Sports Exerc. 2001 Nov;33(11):1841-8. doi: 10.1097/00005768-200111000-00007. PMID 11689733